CLINICAL TRIAL: NCT02655289
Title: Transcutaneous Electrical Nerve Stimulation (TENS) for Advanced Cancer Pain Patients - A Randomized, Double-blind, Placebo-controlled Cross-over Pilot Study
Brief Title: Transcutaneous Electrical Nerve Stimulation (TENS) for Advanced Cancer Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Waldemar Siemens, MSc, University Hospital Freiburg
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: DRKS00007990
Record Dates: First submitted 2016-01-08; First posted 2016-01-14 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modulated TENS (Experimental)
  Interventions: Device: Modulated TENS
- Placebo TENS (Placebo Comparator)
  Interventions: Device: Placebo TENS

INTERVENTIONS:
Device: Modulated TENS — * Frequency: 100 Hz
  * Intensity: individual; TENS should be clearly perceptible but not painful; impulse width is coupled with intensity
  * Mode: intensity modulation (40% decrease every 0.5 seconds)
  * TENS device: ARTROSTIM® SELECT
  * Channels: 2
  * Electrodes: 4 (5x5cm), placed on site of pain (a little more proximal if allodynia is present)
  Arms: Modulated TENS
Device: Placebo TENS — * Frequency: 100 Hz (conventional for High TENS; Placebo is achieved by reduction of intensity, see below)
  * Intensity: The device is on and will be up-regulated together until the first sensation is perceptible. Then the activated device will be down-regulated minimally (no sensation perceptible) and this configuration will be retained.
  * Mode: continuous
  * TENS device: ARTROSTIM® SELECT
  * Channels: 2
  * Electrodes: 4 (5x5cm), placed on site of pain (a little proximal if allodynia is present)
  Arms: Placebo TENS

SUMMARY:
Pain is the most common symptom (ca. 80% of patients) on German Palliative Care units and thus, pain control plays a central role in palliative care.

Transcutaneous electrical nerve stimulation (TENS) is a complementary treatment option for patients who experience suboptimal pain control. However, the evidence for the efficacy of TENS in cancer patients is not unambiguous.

The present study is a double blind, placebo-controlled cross-over trial with a short-term follow-up.

The primary aim of this study is to evaluate the efficacy and safety of TENS for cancer pain reduction in advanced cancer patients.

The secondary aim is the explorative identification of subgroups that benefit or do not benefit from TENS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer pain (caused by tumor or therapy; or associated with tumor) ≥ 3 on an 11-point NRS the last 24 hours
* Age: ≥ 18 years
* Patients receive at least 24 hours palliative care: on palliative care ward, palliative care consultant service or acute pain consultant service

Exclusion Criteria:

* Verbal or cognitive inability to use TENS or to answer the questionnaire
* High probability of dying within the next week
* Pain that is not directly or indirectly related to tumor

Contraindications: Jones (2009) & Disselhoff (2012)

* electronic implants like pacemakers
* Metal implant on electrode site
* Arrhythmia
* Pregnancy
* Epilepsy
* Dermatological conditions or frail skin on electrode site
* Anamnestically known distinct allergy regarding electrodes

Drop-out criteria after inclusion:

* Patients that decide to stop TENS treatment (at any time or any reason).
* Further treatment is not indicated due a rapid deterioration of the patients' clinical status according to the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change of mean pain intensity last 24 hours | Before and after the 24-hour-interventions and after the follow-up: at an average of one week
  11-point Numerical Rating Scale (NRS): 0-10; 0=no pain; 10=pain as bad as you can imagine

SECONDARY OUTCOMES:
Change of worst pain intensity last 24 hours | Before and after the 24-hour-interventions and after the follow-up: at an average of one week
  11-point NRS
Change of least pain intensity last 24 hours | Before and after the 24-hour-interventions and after the follow-up: at an average of one week
  11-point NRS
Change of pain perception during TENS application on NRS | After the 24-hour-interventions and after the follow-up: at an average of one week
  11-point NRS 0-100%; 0% = no alleviation, 100% = complete alleviation
Change of pain perception during TENS application on VRS | After the 24-hour-interventions and after the follow-up: at an average of one week
  7-point verbal rating scale (VRS): 1= "very considerable deterioration", 2= "considerable deterioration", 3= "slight deterioration", 4= "unchanged", 5="slight improvement", 6= "considerable improvement", 7= "very considerable improvement"
Number and percent of responders | After the 24-hour-interventions and after the follow-up: at an average of one week
  Responders: Patients with at least "slight improvement" on VRS (see outcome before) during TENS application
Quality of life last 24 hours | Before and after the 24-hour-interventions and after the follow-up: at an average of one week
  Question 30 from EORTC QLQ-C30
General Activity | Before and after the 24-hour-interventions and after the follow-up: at an average of one week
  11-point NRS
Mood | Before and after the 24-hour-interventions and after the follow-up: at an average of one week
  11-point NRS
Walking ability | Before and after the 24-hour-interventions and after the follow-up: at an average of one week
  11-point NRS
Normal Work (includes both work outside the home and housework) | Before and after the 24-hour-interventions and after the follow-up: at an average of one week
  11-point NRS
Relations with other people | Before and after the 24-hour-interventions and after the follow-up: at an average of one week
  11-point NRS
Sleep | Before and after the 24-hour-interventions and after the follow-up: at an average of one week
  11-point NRS
Enjoyment of life | Before and after the 24-hour-interventions and after the follow-up: at an average of one week
  11-point NRS

CONTACTS AND LOCATIONS:
Overall Officials: Gerhild Becker, Prof., MD, MA, MSc, Study Chair — University Medical Center Freiburg
Locations (1):
- Clinic for Palliative Care, Medical Center, University of Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Radbruch L, Nauck F, Ostgathe C, Elsner F, Bausewein C, Fuchs M, Lindena G, Neuwohner K, Schulenberg D. What are the problems in palliative care? Results from a representative survey. Support Care Cancer. 2003 Jul;11(7):442-51. doi: 10.1007/s00520-003-0472-6. Epub 2003 May 28. PMID 12774219
- [Background] Hurlow A, Bennett MI, Robb KA, Johnson MI, Simpson KH, Oxberry SG. Transcutaneous electric nerve stimulation (TENS) for cancer pain in adults. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD006276. doi: 10.1002/14651858.CD006276.pub3. PMID 22419313
- [Background] Bennett MI, Hughes N, Johnson MI. Methodological quality in randomised controlled trials of transcutaneous electric nerve stimulation for pain: low fidelity may explain negative findings. Pain. 2011 Jun;152(6):1226-1232. doi: 10.1016/j.pain.2010.12.009. Epub 2011 Mar 23. PMID 21435786
- [Background] Bennett MI, Johnson MI, Brown SR, Radford H, Brown JM, Searle RD. Feasibility study of Transcutaneous Electrical Nerve Stimulation (TENS) for cancer bone pain. J Pain. 2010 Apr;11(4):351-9. doi: 10.1016/j.jpain.2009.08.002. Epub 2009 Oct 22. PMID 19853518
- See also: Worldwide Palliative Care Alliance: Global Atlas of Palliative Care at the End of Life. — http://www.thewhpca.org/resources/global-atlas-on-end-of-life-care